CLINICAL TRIAL: NCT00405639
Title: To Define in Human Preclinical Systolic Dysfunction (PSD) the Actions of Chronic Administration of Subcutaneous (SQ) BNP on the Left Ventricular, Renal, and Humoral Function and on the Integrated Response to Acute Sodium Loading
Brief Title: Human B-type Natriuretic Peptide (BNP) (Nesiritide) to Help Heart, Kidney, and Hormonal Functions in Persons With Lower Heart Pumping Function
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Horng Chen, Dr Horng H. Chen, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 05-004186; P01HL076611 (NIH); UL1RR024150 (NIH)
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Results first posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-02

CONDITIONS: Heart Failure; Asymptomatic Systolic Dysfunction
MeSH Terms: conditions — Heart Failure | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nesiritide (Active Comparator): Subjects randomized to this arm will receive 5 microgram/Kg subcutaneous (SQ) injection of nesiritide on Day 1. If after the first SQ injection the subject's systolic blood pressure is >90 mmHG and no symptoms of hypotension, then the second dose can be increased to 10 microgram/Kg. Subjects will self-administer the second dose 12 hours after the first dose, then self-administer the third dose 12 hours after the second dose. Subjects will be dismissed with instructions and supplies for 6 weeks of SQ administration twice a day. After 6 weeks, the subjects will return to the lab for assessments, and will be dismissed with supplies for 6 more weeks of SQ administration twice a day.
  Interventions: Drug: Nesiritide
- Placebo (Placebo Comparator): Subjects randomized to this arm will receive self administered SQ placebo (normal saline) injections to match those of the study drug group. That is, first dose on Day 1, second dose 12 hours after the first dose, third dose 12 hours after the second dose. Subjects will be dismissed with instructions and supplies for 6 weeks of SQ administration twice a day. After 6 weeks, the subjects will return to the lab for assessments, and will be dismissed with supplies for 6 more weeks of SQ administration twice a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nesiritide — Subjects randomized to this arm will receive 5 microgram/Kg subcutaneous (SQ) injection of nesiritide on Day 1. If after the first SQ injection the subject's systolic blood pressure is >90 mmHG and no symptoms of hypotension, then the second dose can be increased to 10 microgram/Kg. Subjects will self-administer the second dose 12 hours after the first dose, then self-administer the third dose 12 hours after the second dose. Subjects will be dismissed with instructions and supplies for 6 weeks of SQ administration twice a day. After 6 weeks, the subjects will return to the lab for assessments, and will be dismissed with supplies for 6 more weeks of SQ administration twice a day.
  Other Names: Natrecor; Human B-type natriuretic peptide (BNP)
  Arms: Nesiritide
Drug: Placebo — Normal saline will be used for placebo.
  Arms: Placebo

SUMMARY:
The following are done for screening procedures to determine if patients are eligible for this study: blood count, kidney and liver blood tests. Patients will complete a 6-minute walk test. Patients will be instructed to follow a no-added-salt diet for 1-3 weeks before the study and for the whole duration of the study. Diet instructions will be given to the patient and the patient will collect his/her urine for 24 hours before the active study day. Patients will need to avoid strenuous exercise and abstain from smoking, alcohol, and caffeine for 3 days prior to the study days. Patients will remain on their regular medications.

DETAILED DESCRIPTION:
Participants in this study will be randomized to receive BNP or placebo (an inactive, saline shot). The participant will need to give themselves a shot in their stomach (similar to diabetics giving themselves insulin) twice a day for twelve weeks. The study requires a screening visit to determine eligibility and discuss the study. At this visit a blood draw for heart and liver function and a six minute walk will be done. There will also be two other outpatient visits and two inpatient stays, for 48 hours, in the General Clinical Research Center (GCRC) at St. Marys Hospital. During the two in-patient stays in the GCRC, blood and urine samples will be done to get heart and kidney function as well as a research echo. After enrollment, the study lasts for twelve weeks. There is a one week visit in outpatient setting getting a blood draw and a 6 week visit in outpatient setting to get a blood draw, 24 hour urine collection and resupply the study medication. There is a one week visit in outpatient setting getting a blood draw and a 6 week visit in outpatient setting to get a blood draw, 24 hour urine collection and resupply the study medication.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with an ejection fraction of less than 45%
* No clinical signs or symptoms of congestive heart failure
* Ability to walk a minimal distance of > 450 meters on a 6-minute walk. If the subject is not able to walk 450 meters due to pain in hips and knees and not fatigue or shortness of breath, they will still qualify for the protocol.
* The subjects will all be on stable doses of an angiotensin converting enzyme (ACE) inhibitor for two weeks prior to the active study date.
* Therapy with other vasodilators, beta-receptor antagonists, digoxin and antiarrhythmic medications will be allowed, however, all medications must be at stable doses two weeks prior to the study date.

Exclusion criteria:

* Myocardial infarction within 3 months of screening
* Unstable angina within 14 days of screening, or any evidence of myocardial ischemia
* Significant valvular stenosis, hypertrophic, restrictive or obstructive cardiomyopathy, constrictive pericarditis, primary pulmonary hypertension, or biopsy proven active myocarditis
* Severe congenital heart diseases
* Sustained ventricular tachycardia or ventricular fibrillation within 14 days of screening
* Second or third degree heart block without a permanent cardiac pacemaker
* Stroke within 3 months of screening, or other evidence of significantly compromised central nervous system (CNS) perfusion
* Total bilirubin of > 1.5 mg/dL or other liver enzymes >1.5 times the upper limit of normal
* Serum creatinine of > 3.0 mg/dL
* Serum sodium of < 125 milliequivalent (mEq)/dL or > 160 mEq/dL
* Serum potassium of < 3.5 mEq/dL or > 5.0 mEq/dL change to 5.3
* Serum digoxin level of > 2.0 ng/ml
* Systolic pressure of < 85 mmHg
* Hemoglobin < 10 gm/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-06; Primary Completion 2011-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horng H. Chen, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were recruited from the Mayo Clinic in Rochester, Minnesota.
Period: Overall Study
Arm/Group | Nesiritide | Placebo
Started | 25 | 12
Completed | 22 | 12
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Seizure prior to receiving BNP | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nesiritide | Placebo | Total
Number analyzed (Participants) | 25 | 12 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 8 | 19
  >=65 years | 14 | 4 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 22 | 10 | 32
Region of Enrollment [Number; unit: participants]
  United States | 25 | 12 | 37

OUTCOME MEASURES:

1. Secondary Outcome: Change in Urine Flow in Response to Saline Load
Time Frame: baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Nesiritide | Placebo
Number analyzed (Participants) | 22 | 12
ml/min | 3.1 (3.8) | -0.4 (2.1)
Statistical Analysis 1: Comparison: Nesiritide; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

2. Secondary Outcome: Change in Renal Function as Measured by Glomerular Filtration Rate (GFR) in Response to Saline Load
Description: Kidney function was measured by GFR determined by iothalamate clearance. GFR describes the flow rate of filtered fluid through the kidney measured in milliliters per minute per 1.73 m^2 of body surface area. A lower GFR means the kidney is not filtering normally. An estimated GFR of less than 60 mg/min/1.73 m^2 of body surface area is considered to be impaired kidney function.
Time Frame: baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: ml/min/1.73 m^2
Arm/Group | Nesiritide | Placebo
Number analyzed (Participants) | 22 | 12
ml/min/1.73 m^2 | 1.6 (9.7) | -7.4 (12.5)
Statistical Analysis 1: Comparison: Nesiritide vs Placebo; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

3. Secondary Outcome: Change in Left Ventricular Mass Index
Description: Left ventricular mass index (LVMI) is a surrogate of left ventricular hypertrophy and a predictor of cardiac morbidity and mortality in adults with hypertension. LVMI was measured with echocardiography, indexed to body surface area estimated by left ventricular (LV) cavity dimension and wall thickness at end-diastole.
Time Frame: baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: g/m^2
Arm/Group | Nesiritide | Placebo
Number analyzed (Participants) | 22 | 12
g/m^2 | -5.8 (15.7) | 2.0 (5.4)
Statistical Analysis 1: Comparison: Nesiritide vs Placebo; Test type: Superiority or Other; p = 0.07, t-test, 2 sided

4. Primary Outcome: Change in Urinary Sodium Excretion in Response to Saline Load
Time Frame: baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: mEq/min
Arm/Group | Nesiritide | Placebo
Number analyzed (Participants) | 22 | 12
mEq/min | 179.1 (252.2) | 3.1 (102.4)
Statistical Analysis 1: Comparison: Nesiritide vs Placebo; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Subjects will be followed for the 12 weeks while on study.
Arm/Group | Nesiritide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/12
Other Adverse Events (participants affected / at risk) | 10/22 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nesiritide (N=22) | Placebo (N=12)
Blurring Vision (Eye disorders) | 0 (0) | 1 (1)
Hypotension (Investigations) | 6 (6) | 1 (1)
Flank pain (Nervous system disorders) | 1 (1) | 0 (0)
Gout (General disorders) | 1 (1) | 0 (0)
Heart Failure symptoms (Cardiac disorders) | 2 (2) | 0 (0)
Hyperkalemia (Vascular disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Thromboembolism (Vascular disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Hospitalization (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No